CLINICAL TRIAL: NCT00097955
Title: Safety and Efficacy of Aliskiren When Added to Standardized Losartan and Optimal Antihypertensive Therapy in Patients With Hypertension, Type 2 Diabetes and Proteinuria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CSPP100C2201; NCT00219206 (obsolete NCT alias)
Record Dates: First submitted 2004-12-01; First posted 2004-12-02 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Diabetic Nephropathy
Keywords: diabetes; nephropathy; hypertension; aliskiren; losartan
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus; Kidney Diseases; Hypertension | interventions — aliskiren

INTERVENTIONS:
Drug: aliskiren

SUMMARY:
Study of the efficacy and safety of aliskiren when added to losartan and optimal antihypertensive therapy in patients with hypertension, type 2 diabetes, and kidney disorders to monitor improvement in any of these conditions.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension
* Elevated urinary protein levels
* Confirmed type 2 diabetes

Exclusion Criteria:

* Certain diseases
* Uncontrolled diabetes
* Type 1 diabetes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 496
Dates: Start 2004-10; Primary Completion 2007-04 (Actual); Study Completion 2007-04

PRIMARY OUTCOMES:
Change from baseline in urinary albumin creatinine ratio after 24 weeks

SECONDARY OUTCOMES:
Equal/more than 50% reduction from baseline in urinary albumin creatinine ratio after 24 weeks
Change from baseline in urinary albumin excretion rate after 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States
- Investigative Site, Québec, Canada
- Investigative Site, Hillerød, Denmark
- Investigative Site, Paris, France
- Investigative Centers, Germany
- Investigative Site, Athens, Greece
- Investigative Site, Rome, Italy
- Investigative Site, Rotterdam, Netherlands
- Investigative Site, Bucharest, Romania
- Investigative Site, Moscow, Russia
- Investigative Site, Madrid, Spain
- Investigative Site, London, United Kingdom

REFERENCES:
- [Derived] Persson F, Lewis JB, Lewis EJ, Rossing P, Hollenberg NK, Parving HH; AVOID Study Investigators. Impact of baseline renal function on the efficacy and safety of aliskiren added to losartan in patients with type 2 diabetes and nephropathy. Diabetes Care. 2010 Nov;33(11):2304-9. doi: 10.2337/dc10-0833. Epub 2010 Aug 6. PMID 20693353
- [Derived] Parving HH, Persson F, Lewis JB, Lewis EJ, Hollenberg NK; AVOID Study Investigators. Aliskiren combined with losartan in type 2 diabetes and nephropathy. N Engl J Med. 2008 Jun 5;358(23):2433-46. doi: 10.1056/NEJMoa0708379. PMID 18525041